CLINICAL TRIAL: NCT00979602
Title: A Study to Evaluate the Safety, Immunogenicity, and Relative Efficacy of A/California/7/2009 (H1N1)V-like Vaccines GSK2340274A and GSK2340273A in Adults Aged 18 Years and Older
Brief Title: Safety, Immunogenicity, and Relative Efficacy of H1N1 Vaccines in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113480
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340274A; Influenza Vaccines; GSK Bio's influenza vaccine GSK2340273A; influenza infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK2340274A Group (Experimental): Healthy male or female subjects between and including 18 to 60 years of age and older (>60 years) and between 18 to 64 years of age and older (>64 years), who received one dose of the adjuvanted GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK2340274A
- GSK2340273A Group (Experimental): Healthy male or female subjects between and including 18 to 60 years of age and older (>60 years) and between 18 to 64 years of age and older (>64 years), who received one dose of the unadjuvanted GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK2340273A

INTERVENTIONS:
Biological: GSK2340274A — One intramuscular injection
  Arms: GSK2340274A Group
Biological: GSK2340273A — One intramuscular injection
  Arms: GSK2340273A Group

SUMMARY:
The purpose of this study is to characterize the safety, immunogenicity, and relative efficacy of the H1N1 (swine) flu vaccines GSK2340273A and GSK2340274A in adults 18 years of age or older.

DETAILED DESCRIPTION:
Collaborators: United States Department of Health and Human Services, Office of Biomedical Advanced Research and Development Authority

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Male and female adults, >= 18 years of age at the time of the first vaccination.
* Satisfactory baseline medical assessment by history and physical examination.
* Safety laboratory test results within the parameters specified in the protocol.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits as demonstrated by signature on the informed consent document.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination; and
* has a negative pregnancy test on the day of first vaccination; and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Previous vaccination at any time with an A/California/7/2009 (H1N1)v-like virus vaccine.
* With the exception of seasonal influenza vaccination, administration of any vaccine(s) within 30 days before study vaccination on Day 0. Seasonal influenza vaccine may be administered up to 14 days prior to study vaccination on Day 0.
* Planned administration of any vaccine other than the study vaccines between Day 0 and the phlebotomy 21 days after vaccination.
* Planned administration of any monovalent pandemic (H1N1)v-like vaccine other than the study vaccines during the whole study (Day 0 - Day 385).
* Previous vaccination with an H1N1v-like virus vaccine or a medical history of physician-confirmed infection with an H1N1v-like virus.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC (>= 100.4 ºF), oral temperature assessment preferred, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Receipt of systemic glucocorticoids within 1month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors, or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* History of an acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* With the exception of seasonal influenza vaccination, administration of any vaccines within 30 days before study vaccination on Day 0. Seasonal influenza vaccine may be administered up to 14 days prior to study vaccination on Day 0.
* Planned administration of any vaccine other than the study vaccine between Day 0 and the phlebotomy 21 days after the second study vaccine dose.
* Use of any investigational or non-registered product within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to vaccination.
* Lactating or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4048 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2011-01-10 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (24):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Camillus, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Willoughby Hills, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Wenatchee, Washington
- Canada (12):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, St-Romulad, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yang WH, Dionne M, Kyle M, Aggarwal N, Li P, Madariaga M, Godeaux O, Vaughn DW. Long-term immunogenicity of an AS03-adjuvanted influenza A(H1N1)pdm09 vaccine in young and elderly adults: an observer-blind, randomized trial. Vaccine. 2013 Sep 13;31(40):4389-97. doi: 10.1016/j.vaccine.2013.07.007. Epub 2013 Jul 12. PMID 23856331
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113480 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340274A Group | GSK2340273A Group
Started | 2025 | 2023
Completed | 1880 | 1890
Not Completed | 145 | 133
Not completed — Serious Adverse Event | 5 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 31 | 25
Not completed — Lost to Follow-up | 100 | 96
Not completed — Migrated/moved from study area | 3 | 6
Not completed — Others | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340274A Group | GSK2340273A Group | Total
Number analyzed (Participants) | 2025 | 2023 | 4048
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (18.6) | 45.4 (18.3) | 45.5 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1185 | 1185 | 2370
  Male | 840 | 838 | 1678
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 118 | 113 | 231
  Geographic ancestry: American Indian or Alaskan native | 14 | 11 | 25
  Geographic ancestry: Asian - Central/South Asian Heritage | 35 | 42 | 77
  Geographic ancestry: Asian - East Asian Heritage | 13 | 8 | 21
  Geographic ancestry: Asian - Japanese Heritage | 4 | 4 | 8
  Geographic ancestry: Asian - South East Asian Heritage | 8 | 7 | 15
  Geographic ancestry: Native Hawaiian or other Pacific Islander | 1 | 2 | 3
  Geographic ancestry: White - Arabic/North African Heritage | 19 | 24 | 43
  Geographic ancestry: White - Caucasian/European Heritage | 1787 | 1790 | 3577
  Geographic ancestry: Other | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: A seroconverted subject was defined as a vaccinated subject who had a post-vaccination titer higher than or equal to (≥)1:40 or at least a 4-fold increase of the pre-vaccination titer of ≥ 1:10. The Flu strain assessed was A/California/7/09 (H1N1)v-like (Flu A/CAL/7/09) in subjects of 18-60 years and older and 18-64 years and older, following the Committee for Medicinal Products for Human Use (CHMP) and the Center for Biologics Evaluation and Research (CBER) guidance.
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 21, which included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against A/California-like HA antigen for the blood sample taken on Day 21 were available.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340274A (18-60 y) Group: Healthy male or female subjects between and including 18 and 60 years of age, who received one dose of the adjuvanted GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340274A (>60 y) Group: Healthy male or female subjects older than 60 years of age (>60 y), who received one dose of the adjuvanted GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340273A (18-60 y) Group: Healthy male or female subjects between and including 18 and 60 years of age, who received one dose of the unadjuvanted GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340273A (>60 y) Group: Healthy male or female subjects older than 60 years of age (>60 y), who received one dose of the unadjuvanted GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340274A (18-64 y) Group: Healthy male or female subjects between and including 18 and 64 years of age, who received one dose of the adjuvanted GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340274A (>64 y) Group: Healthy male or female subjects older than 64 years of age (>64 y), who received one dose of the adjuvanted GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340273A (18-64 y) Group: Healthy male or female subjects between and including 18 and 64 years of age, who received one dose of the unadjuvanted GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
- GSK2340273A (>64 y) Group: Healthy male or female subjects older than 64 years of age (>64 y), who received one dose of the unadjuvanted GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm.
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1345 | 535 | 1338 | 531 | 1426 | 454 | 1414 | 455
Participants | 1210 | 411 | 1012 | 301 | 1279 | 342 | 1055 | 258

2. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the Flu A/CAL/7/09 H1N1 Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) antibody titer ≥ 1:40 against the tested virus. The Flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 0
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 21, which included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against A/California-like HA antigen for the blood sample taken on Day 21 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1347 | 535 | 1344 | 532 | 1428 | 454 | 1420 | 456
Participants | 337 | 74 | 332 | 92 | 350 | 61 | 346 | 78

3. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the Flu A/CAL/7/09 H1N1 Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum HI antibody titer ≥ 1:40. The Flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1350 | 539 | 1347 | 533 | 1432 | 457 | 1424 | 456
Participants | 1326 | 470 | 1246 | 371 | 1403 | 393 | 1302 | 315

4. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: SCF was defined as the fold increase in serum HI geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus, in subjects 18-60 years and older and 18-64 years and older, following the CHMP guidance.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1345 | 535 | 1338 | 531 | 1426 | 454 | 1414 | 455
Fold increase | 27.7 [25.7 to 29.9] | 12.5 [11.2 to 13.9] | 15.5 [14.2 to 16.8] | 6.4 [5.7 to 7.1] | 26.9 [25.0 to 29.0] | 11.9 [10.5 to 13.4] | 14.8 [13.6 to 16.1] | 6.3 [5.5 to 7.1]

5. Primary Outcome: Number of A/California/7/2009 (H1N1)V-like Illness (ILI) Cases
Description: The analysis focused on Quantitative Reverse Transcription Polymerase Chain Reaction Assay (RT-qPCR)-confirmed A/California/7/2009 (H1N1)v-like illness (ILI) cases.
Time Frame: From Day 14 post-vaccination up to study end (at Day 385)
Population: The analysis was performed on the ATP cohort for efficacy, which included all eligible subjects who received the study vaccine according to their treatment assignment and who were successfully contacted at least once during the active influenza surveillance period after completing the Day 21 study visit.
Measure: Number; unit: Events
Arm/Group | GSK2340274A Group | GSK2340273A Group
Number analyzed (Participants) | 1949 | 1958
Events | 1 | 2

6. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: Cut-off values assessed were greater than or equal to (≥) 1:10 in the sera of subjects seronegative before vaccination.
  The Flu strains assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Days 0 and 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1350 | 539 | 1347 | 533 | 1432 | 457 | 1424 | 456
Participants
  Flu A/CAL/7/09, Day 0: number analyzed (Participants) | 1347 | 535 | 1344 | 532 | 1428 | 454 | 1420 | 456
  Flu A/CAL/7/09, Day 0 | 754 | 293 | 731 | 312 | 803 | 244 | 775 | 268
  Flu A/CAL/7/09, Day 21 | 1348 | 534 | 1335 | 512 | 1430 | 452 | 1410 | 437

7. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). The flu strain assessed was /California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Days 0 and 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1350 | 539 | 1347 | 533 | 1432 | 457 | 1424 | 456
Titers
  Flu A/CAL/7/09, Day 0: number analyzed (Participants) | 1347 | 535 | 1344 | 532 | 1428 | 454 | 1420 | 456
  Flu A/CAL/7/09, Day 0 | 14.9 [13.9 to 16.0] | 11.0 [10.1 to 11.9] | 14.8 [13.8 to 15.8] | 12.2 [11.2 to 13.3] | 14.7 [13.8 to 15.7] | 10.9 [10.0 to 11.9] | 14.7 [13.7 to 15.7] | 12.0 [11.0 to 13.2]
  Flu A/CAL/7/09, Day 21 | 415.0 [391.4 to 440.0] | 135.9 [122.1 to 151.1] | 228.7 [213.5 to 245.0] | 77.3 [68.4 to 87.4] | 396.2 [373.8 to 419.9] | 128.6 [114.6 to 144.3] | 217.6 [203.3 to 232.9] | 75.2 [65.9 to 85.9]

8. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: Cut-off values assessed were greater than or equal to (≥) 1:10 in the sera of subjects seronegative before vaccination. The Flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 42
Population: The analysis was performed on a subset from the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against A/California-like HA antigen for the blood sample taken on Day 42 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 50 | 50 | 44 | 48 | 52 | 48 | 46 | 46
Participants | 50 | 50 | 44 | 45 | 52 | 48 | 46 | 43

9. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). The flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 42
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 50 | 50 | 44 | 48 | 52 | 48 | 46 | 46
Titers | 288.5 [215.9 to 385.5] | 105.4 [70.8 to 157.0] | 177.2 [121.3 to 259.0] | 47.9 [33.1 to 69.2] | 276.5 [207.1 to 369.0] | 105.9 [70.2 to 159.9] | 170.0 [117.7 to 245.4] | 47.2 [32.1 to 69.3]

10. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: Cut-off values assessed were greater than or equal to ≥ 1:10 in the sera of subjects seronegative before vaccination. The Flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) in subjects 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 182, which included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against A/California-like HA antigen for the blood sample taken on Day 182 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1306 | 543 | 1314 | 536 | 1388 | 461 | 1391 | 459
Participants | 1282 | 501 | 1257 | 449 | 1361 | 422 | 1324 | 382

11. Secondary Outcome: Titers for Serum HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: as for outcome 9
Time Frame: At Day 182
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1306 | 543 | 1314 | 536 | 1388 | 461 | 1391 | 459
Titers | 115.5 [107.8 to 123.7] | 38.4 [34.6 to 42.6] | 87.6 [81.4 to 94.3] | 30.1 [26.9 to 33.6] | 109.5 [102.3 to 117.1] | 37.1 [33.2 to 41.5] | 83.3 [77.5 to 89.5] | 29.2 [26.0 to 33.0]

12. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: A seroconverted subject was defined as a vaccinated subject who had a post-vaccination titer ≥1:40 and at least a 4-fold increase of the pre-vaccination titer. The Flu strain assessed was A/California/7/09 (H1N1)v-like) (Flu A/CAL/7/09) in subjects of 18-60 years and older and 18-64 years and older, following the CHMP and the CBER guidance.
Time Frame: At Day 42
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 50 | 50 | 44 | 48 | 52 | 48 | 46 | 46
Participants | 49 | 36 | 35 | 20 | 51 | 34 | 36 | 19

13. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: as for outcome 12
Time Frame: At Day 182
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1302 | 539 | 1304 | 534 | 1383 | 458 | 1380 | 458
Participants | 823 | 198 | 717 | 146 | 861 | 160 | 741 | 122

14. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the Flu A/CAL/7/09 H1N1 Virus Strain
Description: as for outcome 3
Time Frame: At Day 42
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 50 | 50 | 44 | 48 | 52 | 48 | 46 | 46
Participants | 49 | 38 | 41 | 29 | 51 | 36 | 43 | 27

15. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the Flu A/CAL/7/09 H1N1 Virus Strain
Description: as for outcome 3
Time Frame: At Day 182
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1306 | 543 | 1314 | 536 | 1388 | 461 | 1391 | 459
Participants | 1091 | 286 | 1009 | 236 | 1140 | 237 | 1047 | 198

16. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 H1N1 Virus Strain
Description: SCF was defined as the fold increase in serum HI geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus, in subjects 18-60 years and older and 18-64 years and older, following the CHMP.
Time Frame: At Day 42
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 50 | 50 | 44 | 48 | 52 | 48 | 46 | 46
Fold increase | 26.8 [20.0 to 35.8] | 11.1 [7.7 to 16.0] | 13.7 [9.1 to 20.6] | 4.0 [2.9 to 5.5] | 26.1 [19.7 to 34.6] | 11.0 [7.5 to 16.1] | 13.2 [8.8 to 19.7] | 3.9 [2.9 to 5.4]

17. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against A/CAL/7/09 H1N1 Virus Strain
Description: as for outcome 16
Time Frame: At Day 182
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A (18-60 y) Group | GSK2340274A (>60 y) Group | GSK2340273A (18-60 y) Group | GSK2340273A (>60 y) Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1302 | 539 | 1304 | 534 | 1383 | 458 | 1380 | 458
Fold increase | 7.7 [7.2 to 8.4] | 3.5 [3.2 to 3.9] | 5.9 [5.4 to 6.4] | 2.5 [2.3 to 2.8] | 7.5 [6.9 to 8.1] | 3.4 [3.0 to 3.8] | 5.6 [5.2 to 6.1] | 2.5 [2.2 to 2.8]

18. Secondary Outcome: Number of A/California Influenza Related Cases
Description: Influenza related cases included: A/California/7/2009 (H1N1)v-like influenza illness (ILI) cases, pneumonia cases, RT-qPCR confirmed influenza, culture confirmed influenza and RT-qPCR confirmed influenza with pneumonia.
Time Frame: From Day 0 up to the end of ILI surveillance (Day 385)
Population: as for outcome 5
Measure: Number; unit: Events
Arm/Group | GSK2340274A Group | GSK2340273A Group
Number analyzed (Participants) | 1949 | 1958
Events
  ILI cases | 195 | 234
  Pneumonia cases | 8 | 21
  RT-qPCR confirmed influenza | 1 | 2
  Culture confirmed influenza | 1 | 2
  RT-qPCR confirmed influenza with pneumonia | 0 | 0

19. Secondary Outcome: Number of ILI Symptoms in All Reported ILI Cases
Description: Assessed ILI symptoms were fever [defined as oral temperature equal to or above (≥) 38.5 degrees Celsius (°C)], myalgia (muscle aches all over the body), cough, sore throat, runny/stuffy nose, short of breath, headache, vomiting, diarrhea, chills, fatigue.
Time Frame: From Day 0 up to the end of ILI surveillance (Day 385)
Population: as for outcome 5
Measure: Number; unit: Events
Arm/Group | GSK2340274A Group | GSK2340273A Group
Number analyzed (Participants) | 1949 | 1958
Events
  Fever | 47 | 58
  Myalgia | 109 | 140
  Cough | 104 | 138
  Sore throat | 98 | 140
  Runny or stuffy nose | 103 | 132
  Short of breath | 48 | 54
  Headache | 97 | 134
  Vomiting | 23 | 20
  Diarrhea | 30 | 35
  Chills | 80 | 104
  Fatigue | 106 | 146

20. Secondary Outcome: Number of ILI Symptoms in All Reported ILI Cases
Description: as for outcome 19
Time Frame: From Day 14 post-vaccination through the end of ILI surveillance (Day 385)
Population: as for outcome 5
Measure: Number; unit: Events
Arm/Group | GSK2340274A Group | GSK2340273A Group
Number analyzed (Participants) | 1949 | 1958
Events
  Fever | 45 | 51
  Myalgia | 104 | 128
  Cough | 99 | 127
  Sore throat | 93 | 129
  Runny or stuffy nose | 99 | 119
  Short of breath | 46 | 50
  Headache | 93 | 122
  Vomiting | 21 | 16
  Diarrhea | 28 | 32
  Chills | 76 | 96
  Fatigue | 102 | 132

21. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1529 | 480 | 1531 | 479
Participants
  Any Pain | 1256 | 272 | 458 | 45
  Grade 3 Pain | 55 | 2 | 4 | 0
  Any Redness | 89 | 25 | 11 | 6
  Grade 3 Redness | 0 | 2 | 0 | 0
  Any Swelling | 137 | 28 | 10 | 3
  Grade 3 Swelling | 1 | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 38.0 degrees Celsius (°C)], headache, joint pain at other location, muscle aches, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1529 | 480 | 1531 | 479
Participants
  Any Fatigue | 473 | 84 | 361 | 59
  Grade 3 Fatigue | 23 | 3 | 18 | 0
  Related Fatigue | 382 | 63 | 298 | 48
  Any Headache | 452 | 73 | 421 | 55
  Grade 3 Headache | 24 | 1 | 14 | 1
  Related Headache | 359 | 53 | 312 | 43
  Any Joint pain | 242 | 52 | 135 | 27
  Grade 3 Joint pain | 16 | 3 | 6 | 2
  Related Joint pain | 205 | 43 | 112 | 23
  Any Muscle aches | 600 | 93 | 281 | 35
  Grade 3 Muscle aches | 25 | 4 | 9 | 1
  Related Muscle aches | 531 | 79 | 240 | 26
  Any Shivering | 157 | 23 | 94 | 17
  Grade 3 Shivering | 12 | 1 | 7 | 0
  Related Shivering | 130 | 17 | 76 | 14
  Any Sweating | 106 | 10 | 76 | 6
  Grade 3 Sweating | 4 | 0 | 3 | 0
  Related Sweating | 81 | 7 | 59 | 5
  Any Temperature | 19 | 4 | 16 | 2
  Grade 3 Temperature | 1 | 0 | 0 | 0
  Related Temperature | 7 | 3 | 7 | 0

23. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], alkaline phosphatase [AP], aspartate aminotransferase [AST], basophils [BAS], total bilirubin [T/BIL], bilirubin direct [BIL/D], creatinine [CREA], eosinophils [EOS], hematocrit [HEM], haemoglobin [Hgb], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelets [PLA], red blood cells [RBC], blood urea nitrogen [BUN] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed with respect to normal laboratory values were - unknown, below, within and above for subjects aged 18-64 years (18-64y) and >64 years old (>64y).
Time Frame: At Days 7 and 21
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1527 | 479 | 1524 | 478
Participants
  ALT, Day 7: Unknown | 3 | 1 | 5 | 3
  ALT, Day 7: Below | 0 | 0 | 0 | 0
  ALT, Day 7: Within | 1497 | 471 | 1482 | 472
  ALT, Day 7: Above | 27 | 7 | 37 | 3
  ALT, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  ALT, Day 21: Unknown | 9 | 0 | 4 | 1
  ALT, Day 21: Below | 0 | 0 | 0 | 0
  ALT, Day 21: Within | 1455 | 469 | 1437 | 469
  ALT, Day 21: Above | 29 | 4 | 51 | 4
  AP, Day 7: number analyzed (Participants) | 1527 | 479 | 1523 | 478
  AP, Day 7: Unknown | 3 | 1 | 5 | 3
  AP, Day 7: Below | 1 | 0 | 0 | 0
  AP, Day 7: Within | 1497 | 463 | 1495 | 468
  AP, Day 7: Above | 26 | 15 | 23 | 7
  AP, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  AP, Day 21: Unknown | 9 | 0 | 4 | 1
  AP, Day 21: Below | 2 | 0 | 0 | 0
  AP, Day 21: Within | 1461 | 463 | 1469 | 464
  AP, Day 21: Above | 21 | 10 | 19 | 9
  AST, Day 7: Unknown | 12 | 3 | 14 | 4
  AST, Day 7: Below | 0 | 0 | 0 | 0
  AST, Day 7: Within | 1505 | 475 | 1493 | 473
  AST, Day 7: Above | 10 | 1 | 17 | 1
  AST, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  AST, Day 21: Unknown | 14 | 0 | 6 | 4
  AST, Day 21: Below | 0 | 0 | 0 | 0
  AST, Day 21: Within | 1466 | 472 | 1459 | 468
  AST, Day 21: Above | 13 | 1 | 27 | 2
  BAS, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  BAS, Day 7: Unknown | 15 | 8 | 8 | 1
  BAS, Day 7: Below | 0 | 0 | 0 | 0
  BAS, Day 7: Within | 1511 | 471 | 1515 | 477
  BAS, Day 7: Above | 0 | 0 | 0 | 0
  BAS, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  BAS, Day 21: Unknown | 35 | 10 | 32 | 8
  BAS, Day 21: Below | 0 | 0 | 0 | 0
  BAS, Day 21: Within | 1458 | 463 | 1460 | 466
  BAS, Day 21: Above | 0 | 0 | 0 | 0
  T/BIL, Day 7: Unknown | 3 | 1 | 5 | 3
  T/BIL, Day 7: Below | 0 | 0 | 0 | 0
  T/BIL, Day 7: Within | 1511 | 475 | 1500 | 472
  T/BIL, Day 7: Above | 13 | 3 | 19 | 3
  T/BIL, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  T/BIL, Day 21: Unknown | 9 | 0 | 4 | 1
  T/BIL, Day 21: Below | 0 | 0 | 0 | 0
  T/BIL, Day 21: Within | 1467 | 468 | 1466 | 467
  T/BIL, Day 21: Above | 17 | 5 | 22 | 6
  BIL/D, Day 7: Unknown | 3 | 1 | 5 | 3
  BIL/D, Day 7: Below | 0 | 0 | 0 | 0
  BIL/D, Day 7: Within | 1524 | 478 | 1518 | 475
  BIL/D, Day 7: Above | 0 | 0 | 1 | 0
  BIL/D, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  BIL/D, Day 21: Unknown | 9 | 0 | 4 | 1
  BIL/D, Day 21: Below | 0 | 0 | 0 | 0
  BIL/D, Day 21: Within | 1484 | 473 | 1488 | 473
  BIL/D, Day 21: Above | 0 | 0 | 0 | 0
  CREA, Day 7: number analyzed (Participants) | 1527 | 479 | 1523 | 478
  CREA, Day 7: Unknown | 3 | 1 | 5 | 3
  CREA, Day 7: Below | 149 | 35 | 144 | 30
  CREA, Day 7: Within | 1365 | 443 | 1363 | 443
  CREA, Day 7: Above | 10 | 0 | 11 | 2
  CREA, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  CREA, Day 21: Unknown | 9 | 0 | 3 | 1
  CREA, Day 21: Below | 150 | 37 | 136 | 32
  CREA, Day 21: Within | 1324 | 431 | 1345 | 438
  CREA, Day 21: Above | 10 | 5 | 8 | 3
  EOS, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  EOS, Day 7: Unknown | 15 | 8 | 8 | 1
  EOS, Day 7: Below | 64 | 12 | 66 | 10
  EOS, Day 7: Within | 1411 | 437 | 1414 | 449
  EOS, Day 7: Above | 36 | 22 | 35 | 18
  EOS, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  EOS, Day 21: Unknown | 35 | 10 | 32 | 8
  EOS, Day 21: Below | 63 | 20 | 60 | 16
  EOS, Day 21: Within | 1345 | 427 | 1361 | 437
  EOS, Day 21: Above | 50 | 16 | 39 | 13
  HEM, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  HEM, Day 7: Unknown | 13 | 6 | 8 | 1
  HEM, Day 7: Below | 72 | 7 | 82 | 6
  HEM, Day 7: Within | 1429 | 463 | 1416 | 467
  HEM, Day 7: Above | 12 | 3 | 17 | 4
  HEM, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  HEM, Day 21: Unknown | 29 | 9 | 29 | 8
  HEM, Day 21: Below | 88 | 10 | 91 | 9
  HEM, Day 21: Within | 1368 | 451 | 1362 | 453
  HEM, Day 21: Above | 8 | 3 | 10 | 4
  HgB, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  HgB, Day 7: Unknown | 13 | 6 | 8 | 1
  HgB, Day 7: Below | 47 | 4 | 65 | 3
  HgB, Day 7: Within | 1455 | 465 | 1436 | 470
  HgB, Day 7: Above | 11 | 4 | 14 | 4
  HgB, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  HgB, Day 21: Unknown | 29 | 9 | 28 | 8
  HgB, Day 21: Below | 58 | 3 | 68 | 6
  HgB, Day 21: Within | 1399 | 460 | 1385 | 456
  HgB, Day 21: Above | 7 | 1 | 11 | 4
  LYM, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  LYM, Day 7: Unknown | 15 | 8 | 8 | 1
  LYM, Day 7: Below | 5 | 5 | 7 | 7
  LYM, Day 7: Within | 1494 | 466 | 1500 | 468
  LYM, Day 7: Above | 12 | 0 | 8 | 2
  LYM, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  LYM, Day 21: Unknown | 35 | 10 | 32 | 8
  LYM, Day 21: Below | 7 | 7 | 2 | 8
  LYM, Day 21: Within | 1445 | 454 | 1444 | 452
  LYM, Day 21: Above | 6 | 2 | 14 | 6
  MON, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  MON, Day 7: Unknown | 15 | 8 | 8 | 1
  MON, Day 7: Below | 306 | 54 | 290 | 52
  MON, Day 7: Within | 1205 | 417 | 1224 | 423
  MON, Day 7: Above | 0 | 0 | 1 | 2
  MON, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  MON, Day 21: Unknown | 35 | 10 | 32 | 8
  MON, Day 21: Below | 309 | 58 | 304 | 64
  MON, Day 21: Within | 1149 | 404 | 1155 | 402
  MON, Day 21: Above | 0 | 1 | 1 | 0
  NEU, Day 7: number analyzed (Participants) | 1522 | 477 | 1522 | 475
  NEU, Day 7: Unknown | 15 | 8 | 8 | 1
  NEU, Day 7: Below | 42 | 9 | 39 | 11
  NEU, Day 7: Within | 1449 | 454 | 1448 | 459
  NEU, Day 7: Above | 16 | 6 | 27 | 4
  NEU, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  NEU, Day 21: Unknown | 35 | 10 | 32 | 8
  NEU, Day 21: Below | 48 | 18 | 53 | 12
  NEU, Day 21: Within | 1392 | 440 | 1392 | 448
  NEU, Day 21: Above | 18 | 5 | 15 | 6
  PLA, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  PLA, Day 7: Unknown | 15 | 8 | 8 | 2
  PLA, Day 7: Below | 6 | 5 | 8 | 7
  PLA, Day 7: Within | 1498 | 465 | 1501 | 467
  PLA, Day 7: Above | 7 | 1 | 6 | 2
  PLA, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  PLA, Day 21: Unknown | 30 | 11 | 29 | 10
  PLA, Day 21: Below | 7 | 5 | 11 | 6
  PLA, Day 21: Within | 1454 | 456 | 1448 | 456
  PLA, Day 21: Above | 2 | 1 | 4 | 2
  RBC, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  RBC, Day 7: Unknown | 13 | 6 | 8 | 1
  RBC, Day 7: Below | 97 | 6 | 102 | 6
  RBC, Day 7: Within | 1411 | 463 | 1402 | 469
  RBC, Day 7: Above | 5 | 4 | 11 | 2
  RBC, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  RBC, Day 21: Unknown | 29 | 9 | 29 | 8
  RBC, Day 21: Below | 95 | 8 | 90 | 8
  RBC, Day 21: Within | 1368 | 455 | 1367 | 458
  RBC, Day 21: Above | 1 | 1 | 6 | 0
  BUN, Day 7: number analyzed (Participants) | 1527 | 479 | 1523 | 478
  BUN, Day 7: Unknown | 3 | 1 | 5 | 3
  BUN, Day 7: Below | 5 | 0 | 9 | 0
  BUN, Day 7: Within | 1509 | 471 | 1500 | 466
  BUN, Day 7: Above | 10 | 7 | 9 | 9
  BUN, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  BUN, Day 21: Unknown | 9 | 0 | 4 | 1
  BUN, Day 21: Below | 9 | 0 | 5 | 0
  BUN, Day 21: Within | 1462 | 467 | 1467 | 469
  BUN, Day 21: Above | 13 | 6 | 16 | 4
  WBC, Day 7: number analyzed (Participants) | 1526 | 479 | 1523 | 478
  WBC, Day 7: Unknown | 15 | 8 | 8 | 1
  WBC, Day 7: Below | 27 | 10 | 30 | 12
  WBC, Day 7: Within | 1457 | 455 | 1440 | 458
  WBC, Day 7: Above | 27 | 6 | 45 | 7
  WBC, Day 21: number analyzed (Participants) | 1493 | 473 | 1492 | 474
  WBC, Day 21: Unknown | 35 | 10 | 32 | 8
  WBC, Day 21: Below | 31 | 11 | 30 | 10
  WBC, Day 21: Within | 1406 | 448 | 1398 | 444
  WBC, Day 21: Above | 21 | 4 | 32 | 12

24. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1544 | 481 | 1543 | 480
Participants | 615 | 247 | 614 | 265

25. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) represent a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1544 | 481 | 1543 | 480
Participants | 2 | 3 | 4 | 3

26. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: Within the 42-day (Days 0-41) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1544 | 481 | 1543 | 480
Participants | 495 | 119 | 522 | 139

27. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Safety results were tabulated according to age stratification: adults aged 18-64 years and older (>64y).
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A (18-64 y) Group | GSK2340274A (>64 y) Group | GSK2340273A (18-64 y) Group | GSK2340273A (>64 y) Group
Number analyzed (Participants) | 1544 | 481 | 1543 | 480
Participants | 45 | 39 | 32 | 41

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period. Unsolicited AEs: during the 42-day (Days 0-41) post-vaccination period. Serious adverse events (SAE): during the entire study period (Day 0 to Day 385).
Arm/Group | GSK2340274A Group | GSK2340273A Group
All-Cause Mortality (participants affected / at risk) | 6/2025 | 1/2023
Serious Adverse Events (participants affected / at risk) | 84/2025 | 73/2023
Other Adverse Events (participants affected / at risk) | 1680/2025 | 1063/2023
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340274A Group (N=2025) | GSK2340273A Group (N=2023)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Histoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (3)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram st segment elevation (Investigations) | 1 (1) | 0 (0)
Enzyme activity decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicle centre lymphoma, follicular grade i, ii, iii stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340274A Group (N=2025) | GSK2340273A Group (N=2023)
Arthralgia (Musculoskeletal and connective tissue disorders) | 299 (302) | 165 (167)
Chills (General disorders) | 181 (183) | 116 (116)
Cough (Respiratory, thoracic and mediastinal disorders) | 78 (82) | 110 (112)
Erythema (Skin and subcutaneous tissue disorders) | 114 (114) | 18 (18)
Fatigue (General disorders) | 564 (573) | 428 (435)
Headache (Nervous system disorders) | 547 (570) | 510 (530)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 116 (116) | 83 (83)
Myalgia (Musculoskeletal and connective tissue disorders) | 698 (709) | 326 (329)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 122 (124) | 126 (131)
Pain (General disorders) | 1530 (1533) | 508 (509)
Swelling (General disorders) | 165 (165) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.